CLINICAL TRIAL: NCT01439906
Title: Evaluation of Pain Relief and Functional Improvement After the Surgical Treatment for Low Back Pain Due to Degenerative Kyphoscoliosis - Pilot Study
Brief Title: Surgical Treatment for Degenerative Scoliosis
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: CVOD.SCOLIOSI DEGENERATIVA
Record Dates: First submitted 2011-09-21; First posted 2011-09-23 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2014-09

CONDITIONS: Scoliosis; Kyphoscoliosis
Keywords: Degenerative scoliosis; Pain; Deformity correction; Instrumented arthrodesis
MeSH Terms: conditions — Scoliosis; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adult degenerative scoliosis: Patients aged 40-75 years affected by lumbar or thoraco-lumbar degenerative kyphoscoliosis presenting chronic low back pain from six months at least and/or neurological deficits who underwent a surgical correction of the deformity
  Interventions: Procedure: Surgical correction of the deformity

INTERVENTIONS:
Procedure: Surgical correction of the deformity — Three different surgical techniques are used:
  * lumbar fusion vs thoraco-lumbar fusion
  * iliac fixation vs fixation to the sacrum
  * posterior + interbody fusion vs posterior interbody fusion

SUMMARY:
The study aims to analyze the surgical treatment of low back pain due to degenerative kyphoscoliosis, already routinely performed on patients treated in Istituto Ortopedico Rizzoli, in terms of reduction of the pain and functional improvement. The comparison of back pain and functional ability before and after the surgical treatment will be performed by administering to the patients specific questionnaires (Visual Analog Score VAS, Oswestry Disability Index ODI, Quality of Life EuroQoL 5D). Questionnaires administration will be matched to a purely objective and radiological assessment according to international guidelines. A psychological analysis will be also performed in order to evaluate co-morbidity from this field, considering that the concept of "shared decision-making" for the therapeutic approach to low back pain requires the evaluation of all these parameters.

ELIGIBILITY:
Inclusion Criteria:

* Female or male
* Age 40-75 years
* Patients capable of understanding and willing
* Lumbar or thoraco-lumbar degenerative kyphoscoliosis
* Chronic low back pain from more than 6 months and/or presence of neurological deficits at lower limbs
* Failure to respond to conservative therapy

Exclusion Criteria:

* Infections in place
* Coagulation deficits
* Serious psychological comorbidity

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2010-01; Primary Completion 2013-12 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change from the baseline clinical status at 1-3-6-12 months after the surgical treatment for degenerative scoliosis. | Before surgery, 1-3-6-12 months after surgery, then annually
  The clinical status of the patients will be evaluated before surgery and at 1-3-6-12 months of follow up (and then annually) by: 1. Visual Analog Scale (VAS); 2. Oswestry Disability Index (ODI); 3. Quality of life (EuroQoL 5D) test.
Change from the baseline radiographic status at 1-3-6-12 months after the surgical treatment for degenerative scoliosis. | Before surgery, 1-3-6-12 months after surgery, then annually
  The correction of the deformity with respect to the pre-operative status will be assessed by anteroposterior, bending and lateral full standing radiographs at 1-3-6-12 months of follow up (and then annually). Flexion/extension radiographs will be taken at 1-3-6-12 months after surgery in order to evaluate fusion and proper positioning of hardware. Successful arthrodesis (fusion) will be also confirmed by CT scan at 1 year.
  Criteria of fusion evaluation:
  1. Fusion certain
  2. Fusion likely
  3. Status uncertain
  4. Pseudo arthrosis likely
  5. Pseudo arthrosis certain
Assessment of the psychological state of the patients before the surgical treatment and at 1-3-6-12 months of follow up. | Before surgery, 1-3-6-12 months after surgery, then annually
  The psychological state of the patients will be evaluate before the surgical treatment and at 1-3-6-12 months after surgery (then annually).
  To evaluate the psychological state of the patients the following questionnaires will be used:
  * STAI to evaluate the anxiety state
  * ZHUNG to evaluate the depressive state

SECONDARY OUTCOMES:
Evaluation of possible surgical complications (hardware failure, neurological damages, re-intervention) during the perioperative period and at 1-3-6-12 months after surgery. | Perioperative, 1-3-6-12 months after surgery, then annually
  Major and minor surgical complications will be recorded and analysed during the perioperative period (early complications) and at 1-3-6-12 months after surgery (late complications).

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Barbanti Brodano, Dr, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy